CLINICAL TRIAL: NCT06838741
Title: Comparison of Effects of Virtual Reality and Otago Exercises on Balance, Gait and Activities of Daily Living in Parkinson's Disease Patients.
Brief Title: Effects of Virtual Reality and Otago Exercises in Parkinson's Disease Patients.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0251
Record Dates: First submitted 2025-01-01; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: Activities of daily living; Balance, gait; otago exercises; Parkinsons disease; Virtual reality
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A Otago exercises (Experimental): It comprises 12 balance exercises and 5 strengthening exercises. The exercises are to be done by participants three times a week. Exercises can be advanced by adding weight or repetitions, contingent on the person's strength and range of motion (weighted ankle cuffs can be utilized and modified during the program).
  Interventions: Procedure: otago exercises; Device: virtual reality
- Group B Virtual reality (Experimental): Participants in this group will receive virtual realityBegin with 20-30 minutes per session and extend to 30-45 minutes as tolerance and endurance improve throughout the program. Exercise sessions will be done for 3 sessions per week.
  Interventions: Procedure: otago exercises; Device: virtual reality

INTERVENTIONS:
Procedure: otago exercises — A walking program is given to participants, with the goal of including two 30-minute walking sessions each week (which can be divided into shorter segments, like three ten-minute blocks).
  Exercises Start exercises with 10 repetition maximum STRENGTH Knee extensor Hold for 3-5 seconds Knee flexor Hold for 3-5 seconds Hip adductor Hold for 3-5 seconds Ankle planter-flexion Calf raises Ankle dorsiflexion Toe raise BALANCE Knee bends Backwards walking Upto 30 minutes Walking and turning around 5-10 minutes Sideways walking Tandem stance Heel to toe stand Tandem walk One leg stand Heel walking Toe walk Heel toe walking backwards Sit to stand Stair walking
Device: virtual reality — Begin with 20-30 minutes per session and extend to 30-45 minutes as tolerance and endurance improve throughout the program. Exercise sessions will be done for 3 sessions per week.

SUMMARY:
Parkinson's disease, the second most common neurological condition, significantly affects motor function, gait, balance, and daily living activities. There is a pressing need for advanced therapies that specifically address these challenges. This study explores the potential benefits of virtual reality and Otago exercises, which may enhance balance and gait by providing sensory feedback crucial for motor learning and relearning. The randomized clinical trial will enroll 74 participants with Parkinson's disease, selected through non-probability convenience sampling. After obtaining synopsis approval, participants will be randomly assigned to one of two groups: Group A will engage in Otago exercises, while Group B will participate in virtual reality sessions. Each treatment session will last for 25 minutes. To evaluate outcomes, various tools will be employed, including the Berg Balance Scale for static balance and the Timed Up and Go test for dynamic balance. The 6-Minute Walk Test will measure gait performance, and the Unified Parkinson Disease Rating Scale will assess activities of daily living. Data normality will be determined using the Kolmogorov-Smirnov test, with subsequent analyses employing either one-way ANOVA or the Kruskal-Wallis test, depending on data distribution, to draw meaningful conclusions regarding treatment efficacy.

DETAILED DESCRIPTION:
The second most prevalent neurological condition is Parkinson disease. It impairs motor function, gait, balance, and daily living tasks. More advanced therapies that target balance, gait, and activities of daily living are required. Virtual reality helps in cognitive and motor improvement by creating a virtual environment. While otago exercise helps to improve balance and coordination and reduce the risk of falls in Parkinson patients. Virtual reality and otago exercises may help to improve balance and gait by providing sensory feedback that will help in motor learning and relearning. This study will compare the effects of virtual reality and otago exercises on balance, gait, and activities of daily living in patients with Parkinson's disease.

This randomized clinical trial will be carried out in a study setting 10 months after the approval of synopsis. In this study, 74 participants who will meet inclusion criteria through a non-probability convenience sampling technique will be included. Participants will be randomly assigned into 2 groups using online research randomizer software. Group A and Group B participants will receive Otago exercises and virtual reality, respectively. Total treatment time will be 25 minutes. The outcome measuring tools used will be Berg balance scale for static balance and time-up and go to measure dynamic balance; a 6-minute walk test will be used for gait, and Unified Parkinson disease Rating scale for activities of daily living. Kolmogorv-Smirnov test will be used to check normality of data. If data will be normally distributed, a one-way ANOVA will be used, and for non-parametric data, the Kruskal-Wallis test will be used.

Type (Exercises):

Weeks 1-2: Foundation and Familiarization Balance Exercises: Start with basic static balance tasks (e.g., standing on one leg, weight shifting) within a VR environment.

Gait preparation: introduce walking simulations on level ground to familiarize participants with VR-based gait training.

ADL Simulation: Initiate simple ADL tasks in VR, such as reaching for objects or virtual button pressing.

Weeks 3-4: Balance and Coordination Development

* Dynamic Balance: Progress to dynamic balance exercises (e.g., stepping over virtual obstacles, balancing on unstable surfaces in VR).
* Coordination Training: Incorporate dual-task activities where participants perform balance exercises while engaging in cognitive tasks within the VR environment.
* Functional ADLs:

ELIGIBILITY:
Inclusion criteria

* The age group of 50 to 70 years will be included (19).
* Both male and female (20) .
* Patients diagnosed with Parkinson's disease of Hoehn and Yahr stage (1-3)
* Patient should be able to stand 10 minutes at least without assistance.
* Patients should be able to walk with or without assistance.
* Mini mental score should be higher than 24

Exclusion Criteria

* Recent surgery or any fracture.
* Any visual and hearing impairments.
* Any pathology that may impair therapy
* Joint pain or musculoskeletal problem that interfered with therapy (22).

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-05-02 (Estimated)

PRIMARY OUTCOMES:
Berg Balance scale | 12 weeks
  It is a 14-item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait. A score of 56 indicates functional balance. A score of < 45 indicates individuals may be at greater risk of falling. A score of ≤49 indicates a risk of falls in individuals with stroke
Time Up and Go test | 12 weeks
  The patient starts in a seated position. The patient stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated. An older adult who takes ≥12 seconds to complete the TUG is at risk for falling. In Parkinson's, the patient is at high risk of fall if he takes more than 11.5 seconds. High test-retest reliability in patients with Parkinson's Disease (ICC= 0.80).
Unified Parkinson Disease Rating Scale (Activities of Daily Living) | 12 weeks
  This part consist of 13 items speech, salivation, swallowing, handwriting, cutting food and handling utensils, dressing, hygiene, turning in bed and changing clothes, falling, freezing while walking, walking, tremor, sensory complains related to parkinsonism. Score ranging from 0-4, higher the score more will be severity.

SECONDARY OUTCOMES:
mini mental scale | 10 minutes
  The MMSE includes tasks that measure various cognitive domains such as orientation, memory, attention, calculation, language, and visuospatial abilities. Typically, the exam takes about 10 minutes to administer and consists of a series of questions and simple tasks. Scoring ranges from 0 to 30, with lower scores indicating greater cognitive impairment. It is commonly used in diagnosing and tracking conditions like dementia and Alzheimer's disease

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, MS, Principal Investigator — Riphah International University
Locations (1):
- General hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yu X, Wu X, Hou G, Han P, Jiang L, Guo Q. The Impact of Tai Chi on Motor Function, Balance, and Quality of Life in Parkinson's Disease: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2021 Jan 11;2021:6637612. doi: 10.1155/2021/6637612. eCollection 2021. PMID 33505498
- [Background] Bloem BR, Okun MS, Klein C. Parkinson's disease. Lancet. 2021 Jun 12;397(10291):2284-2303. doi: 10.1016/S0140-6736(21)00218-X. Epub 2021 Apr 10. PMID 33848468
- [Background] Chua LK, Chung YC, Bellard D, Swan L, Gobreial N, Romano A, Glatt R, Bonaguidi MA, Lee DJ, Jin Y, Liu CY, Fisher BE. Gamified Dual-Task Training for Individuals with Parkinson Disease: An Exploratory Study on Feasibility, Safety, and Efficacy. Int J Environ Res Public Health. 2021 Nov 25;18(23):12384. doi: 10.3390/ijerph182312384. PMID 34886114
- [Background] Balestrino R, Schapira AHV. Parkinson disease. Eur J Neurol. 2020 Jan;27(1):27-42. doi: 10.1111/ene.14108. Epub 2019 Nov 27. PMID 31631455
- [Background] Simon DK, Tanner CM, Brundin P. Parkinson Disease Epidemiology, Pathology, Genetics, and Pathophysiology. Clin Geriatr Med. 2020 Feb;36(1):1-12. doi: 10.1016/j.cger.2019.08.002. Epub 2019 Aug 24. PMID 31733690